CLINICAL TRIAL: NCT02109094
Title: Investigating Markers of Energy Metabolism in the CNS and Periphery in Pregnant Women With Varying Degrees of Insulin Resistance
Brief Title: Investigating Markers of Energy Metabolism in Pregnant Women With Insulin Resistance
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1301011387; R01DK020495-37 (NIH)
Record Dates: First submitted 2014-04-04; First posted 2014-04-09 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Gestational Diabetes; Type 2 Diabetes Mellitus
Keywords: insulin; metabolomics
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urine, cerebrospinal fluid, cord blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant
- Not Pregnant

SUMMARY:
The investigators seek to examine the metabolic changes that occur amongst obese and lean pregnant women with normal glycemic control as well as pregnant women with diabetes mellitus (gestational diabetes and pre-existing type 2 diabetes mellitus) compared to non-pregnant age matched controls. Given the adaptive tendency of the maternal body to use alternative energy sources such as ketones and free fatty acids rather than glucose and to shunt glucose and amino acids to the fetus, the investigators hypothesize that the amino acid and fatty acid profile will be reflective of this adaptive change and that maternal insulin resistance will result in alterations in this pattern in both the plasma and CSF. Furthermore, the investigators also hypothesize that maternal degrees of insulin resistance will also be reflected in CSF hormonal changes.

DETAILED DESCRIPTION:
We seek to investigate for the first time whether CSF branched chain amino acid, free fatty acid, and energy regulatory hormone levels are altered in comparison to plasma levels among pregnant and non-pregnant individuals with varying degrees of insulin resistance. Furthermore, we seek to understand the effects of pregnancy on central and peripheral energy metabolism using metabolomic profiling as well as traditional hormonal measurements in maternal blood, urine, cerebrospinal fluid as well as cord blood.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ages 18-45, pre-pregnancy BMI 18-30 with normal glycemic control scheduled for an elective cesarean delivery at Yale-New Haven Hospital on the Labor and Birth unit
* Pregnant women ages 18-45, pre-pregnancy BMI >30 with normal glycemic control scheduled for an elective cesarean delivery at Yale-New Haven Hospital on the Labor and Birth unit
* Pregnant women ages 18-45 with diabetes (gestational or pre-existing type 2 DM) scheduled for an elective cesarean delivery at Yale-New Haven Hospital on the Labor and Birth unit
* Non-pregnant, non-diabetic women age 18-45 scheduled for lumbar puncture at the Yale-New Haven Hospital Lumbar puncture clinic
* Able to read and understand English at 6th grade level or higher

Exclusion Criteria:

* Medical disorders other than diabetes. Including psychiatric disorders, alcohol abuse, HIV, hepatitis, renal, hepatic disease, heart disease, active systemic infection, malignancy
* Pregnancy related medical problems including preeclampsia
* Major congenital fetal anomalies
* Smoking and illicit drugs (marijuana, cocaine, benzodiazepines, barbituates)
* Use of weight loss supplements or dieting 6 months prior to study.
* Corticosteroid use within 6 months of study.
* Uncontrolled thyroid disease
* Medications other than multivitamin, folic acid, or diabetic medications.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All pregnant subjects will be women recruited from the Women's Center, the high-risk prenatal care unit at Tompkins, Long Wharf and L&D.
  The target population in this study includes pregnant women with pregnancies complicated by gestational diabetes, DM, and uncomplicated controls.
  The Yale New Haven Hospital Lumbar puncture clinic, located in the Yale Physicians Building, is a weekly referral clinic in the department of Neurology. The target population for this study includes non-pregnant women, age greater than 18 who require large volume lumbar puncture for medical purposes such as for symptomatic treatment of pseudotumor cerebri.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Insulin Level (mg/dl) | Baseline (At the time of surgery)
Blood Glucose Level (mmol/L) | Baseline (At the time of surgery)
Plasma Leptin Level | Baseline (At the time of surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sherwin, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States